CLINICAL TRIAL: NCT02777307
Title: Efficacy of Hemopatch in Reducing of Postoperative Bleeding After Laparoscopic Cholecystectomy: Prosective and Multicenter Study
Brief Title: Demonstrate the Effectiveness to Hemopatch in Controlling Postoperative Bleeding After Laparoscopic Cholecistectomy and in Reducing of Morbidity and Postoperative Hospital Stay
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedale Regina Apostolorum (Other)
Collaborators: Azienda Ospedaliera San Gerardo di Monza (Other); San Giuseppe Moscati Hospital (Other); Ospedali Riuniti di Foggia (Other)
Responsible Party: Principal Investigator, A. Liverani, Head of surgery department, Ospedale Regina Apostolorum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 474 bis/DS
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Efficacy of Hemopatch in Controlling of Postoperative Bleeding or Reducing of Postperative Morbidity After Laparoscopic Cholecistectomy
Keywords: Laparoscopic; Cholecistectomy; Collection; Bleeding; reoperation
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemopatch Sealing Hemostat (Experimental)
  Interventions: Other: Hemopatch Sealing Hemostat
- No Hemopatch Sealing Hemostat (No Intervention)

INTERVENTIONS:
Other: Hemopatch Sealing Hemostat — Place of Hemopatch Sealing Hemostat after laparoscopic cholecistectomy
  Arms: Hemopatch Sealing Hemostat

SUMMARY:
Demonstrate the effectiveness to Hemopatch in controlling postoperative bleeding or reducing of postperative fluid collection after laparoscopic cholecistectomy, morbidity and postoperative hospital stay.

DETAILED DESCRIPTION:
Prospective Multicenter Longitudinal and cohort. The sample size of 150 patients was calculated in order to obtain a statistical power adequacy or higher (Type I error - Alpha = 0.05, Type II Error - Beta = 0:20), assuming the 1-day to reduce the postoperative stay with use Hemopatch compared to the control (average stay little 3 +/- 2 days).

Primary endpoint:

- significant reduction in postoperative hospital stay

Secondary endpoints:

* reduction of subhepatic blood liquid volume
* reduction of liver hematoma
* reduction of postooperative complications as deep surgical site
* reduction rates of reoperation
* reduction in readmission rates
* postoperative pain on the VAS scale 1-10.

The results obtained in relation to primary and secondary objectives will be compared with a control group of case-matched.

Inclusion Criteria:

- Between the ages of 18-75 years, calculus of gallbladder (micro- and macro-lithiasis), polyp/neoplasm of gallbladder

Exclusion Criteria:

- Coagulopathies, medication with antiplatelet drugs, ASA > 3, acute cholecystitis, simultaneous calculus of main biliary duct, acute pancreatitis.

The patient will enroll if cholecystectomy is performed laparoscopically, if it is not a complication occurred intraoperative type: iatrogenic enterotomy suture intestinal, iatrogenic lesion of liver parenchyma, bile duct injury. The patient will exclude from the study if one of these intraoperative complication will occur. The patient leaves the protocol if the dissection is done through energy-devices (ultrasound or radiofrequency).

At the end of the laparoscopic cholecstectomy, Hemopatch will be inserted into the peritoneal cavity through the port of 10-12 mm and laid on the cavity of the gallbladder and a drainage will be systematically placed.

It will be given a first-generation cephalosporin antibiotic (one shot).

At 24 hours of VLC a liver ultrasound will be performed and recorded: evaluation of presence of perihepatic fluid, collection or haematoma. It will be noted the volume of drainage which will be removed in first postoperative day. In case of delay removal of drainage, it will be recorded. It will be assessed postoperative pain by VAS scales to 6-12-24 h after surgery. Re-operations and re-hospitalizations will be recorded in prospective data.

Statistical analyzes were performed using the software SPSS for Mac, 22nd edition (SPSS Software, Inc., IL, Chicago). The differences in the distributions will be calculated using the chi-square test or Fisher exact test, depending on the number of cases in the various subgroups and by comparing means (Student t-test, one-way ANOVA test).

The p < 0.1 will be used as the cut-off for statistical significance in the selection of variables of multivariate analysis in order not to drop important potential predictors.

The statistical significance is conventionally defined with p <0.05 in all cases considered.

All eligible patients will be adequately informed and informed consent will be signed. The Study will be conducted according to ethical requirements, following the Declaration of Helsinki, and good clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Gallbladder stone
* Polyp/neoplasm of gallbladder

Exclusion Criteria:

* Coagulopathies,
* Medication with antiplatelet agents
* ASA > 3
* Acute cholecystitis
* Main biliaru duct stone
* Acute pancreatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
significant reduction in postoperative hospital stay | 1 year

SECONDARY OUTCOMES:
reducing of subhepatic volume drainage | 1 year
reducing of liver hematoma | 1 year
reducing of postoperative complications | 1 year
reducing of rates of reoperation | 1 year
reducing of re-hospitalization | 1 year
To assess postoperative pain by the VAS scale 1-10. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Apostolorum Hospital, Albano Laziale, Rome, Italy

REFERENCES:
- [Result] Lewis KM, McKee J, Schiviz A, Bauer A, Wolfsegger M, Goppelt A. Randomized, controlled comparison of advanced hemostatic pads in hepatic surgical models. ISRN Surg. 2014 Mar 4;2014:930803. doi: 10.1155/2014/930803. eCollection 2014. PMID 24729905
- [Result] Lewis KM, Spazierer D, Slezak P, Baumgartner B, Regenbogen J, Gulle H. Swelling, sealing, and hemostatic ability of a novel biomaterial: A polyethylene glycol-coated collagen pad. J Biomater Appl. 2014 Nov;29(5):780-8. doi: 10.1177/0885328214545500. Epub 2014 Aug 1. PMID 25085811
- [Result] Imkamp F, Tolkach Y, Wolters M, Jutzi S, Kramer M, Herrmann T. Initial experiences with the Hemopatch(R) as a hemostatic agent in zero-ischemia partial nephrectomy. World J Urol. 2015 Oct;33(10):1527-34. doi: 10.1007/s00345-014-1404-4. Epub 2014 Sep 20. PMID 25239500
- [Result] Lewis KM, Schiviz A, Hedrich HC, Regenbogen J, Goppelt A. Hemostatic efficacy of a novel, PEG-coated collagen pad in clinically relevant animal models. Int J Surg. 2014;12(9):940-4. doi: 10.1016/j.ijsu.2014.07.017. Epub 2014 Aug 6. PMID 25106082
- [Result] Stokes ME, Ye X, Shah M, Mercaldi K, Reynolds MW, Rupnow MF, Hammond J. Impact of bleeding-related complications and/or blood product transfusions on hospital costs in inpatient surgical patients. BMC Health Serv Res. 2011 May 31;11:135. doi: 10.1186/1472-6963-11-135. PMID 21627788
- [Result] Keus F, Wetterslev J, Gluud C, Gooszen HG, van Laarhoven CJ. Trial sequential analyses of meta-analyses of complications in laparoscopic vs. small-incision cholecystectomy: more randomized patients are needed. J Clin Epidemiol. 2010 Mar;63(3):246-56. doi: 10.1016/j.jclinepi.2009.08.023. Epub 2009 Dec 11. PMID 20004553